CLINICAL TRIAL: NCT06243913
Title: Analysis of Reproductive Outcomes Obtained in Patients Undergoing Intrauterine Insemination with Donor Sperm Previously Vitrified - Pilot Study
Brief Title: A Pilot Study Analyzing Reproductive Results After IUI Using Vitrified Human Sperm
Acronym: BIOKIBANK
Status: Completed | Type: Observational
Sponsor: Clínica EUGIN (Other)
Responsible Party: Sponsor
Other Study IDs: BIOKIBANK
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Infertility
Keywords: intrauterine insemination; sperm cryopreservation; sperm vitrification
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention arm: Use of vitrified donor semen for Intrauterine Artificial Insemination
  Interventions: Procedure: IUI with vitrified sperm from donor:

INTERVENTIONS:
Procedure: IUI with vitrified sperm from donor: — After signing the informed consent, the clinic's Matching team will assign a donor semen straw based on phenotypic characteristics, blood group, and genetic compatibility (if applicable), with the female partner.
  On the day of the Intrauterine Insemination (IUI), the laboratory team will thaw the assigned donor semen straw and post-thaw sperm parameters will be analyzed, including the total number of sperm with progressive motility. Subsequently, the IUI will be performed following the standard protocol.

SUMMARY:
The aim of this study is to assess the evaluate the effectiveness of vitrified donor semen in intrauterine insemination treatments.

DETAILED DESCRIPTION:
Sperm cryopreservation is an efficient procedure widely used in fertility clinics, that provides logistical flexibility and increases the potential for success in assisted reproduction. It has been demonstrated that reproductive rates are comparable when using frozen sperm or fresh semen. However, sperm freezing using standard protocols is inevitably associated with a loss of motility, membrane integrity, and other post-thaw sperm quality parameters due to what is known as cryodamage, which involves the formation of intracellular ice crystals, osmotic shock, and dehydration.

Sperm vitrification has been recently developed as an improved alternative, where freezing occurs extremely rapidly (-20,000 ºC/min). Consequently, the formation of intracellular ice crystals is reduced, leading to improvements in sperm motility, vitality, and integrity.

However, the use of vitrified semen in fertility clinics is scarce, and no study has addressed whether vitrification could affect reproductive outcomes, such as live birth.

The aim of this study is to assess the evaluate the effectiveness of vitrified donor semen in intrauterine insemination treatments through the analysis of clinical pregnancy (primary objective) and as secondary objectives the number of progressive sperm post-thaw, percentage of progressive sperm and biochemical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Artificial Insemination with sperm from donor.
* Female partner's age < 35 years
* First IUI attempt
* Caucasian phenotype

Exclusion Criteria:

* Any adverse medical condition that may significantly affect reproductive outcomes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ART couples where the female partner is under 35 years old who are undergoing their first attempt of intrauterine artificial insemination with donor semen
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks after procedure
  Fetal heartbeat observed in the 7th week of gestation.

SECONDARY OUTCOMES:
Percentage of sperm progressive motility | Day of procedure
  Percentage of sperm progressive motility (% a+b) after thawing
Total number of sperm with progressive motility | Day of procedure
  Total number of sperm with progressive motility after thawing
Biochemical pregnancy rate | 14 days after procedure
  Positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Marc Torra-Massana, PhD, Principal Investigator — Clinica EUGIN, Barcelona (Spain)
Locations (1):
- Clinica EUGIN, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No